CLINICAL TRIAL: NCT05645562
Title: Effects of the Pain Education Program in the Sport Population
Brief Title: Pain Education Program in the Sport Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 280CER22
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2023-03

CONDITIONS: Pain; Sports; Education
Keywords: Pain education; Athlete; Pain catastrophizing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will receive a pain neuroscience education program (once time per month, during 4 months). This program will include information about biological, psychological and perceptual aspects of pain in the sport context.
  Interventions: Behavioral: Pain neuroscience education program
- Control group (Active Comparator): The control group will receive a self-care education program (once time per month, during 4 months). This program will include information about health habits in the sport.
  Interventions: Behavioral: Self-care education program

INTERVENTIONS:
Behavioral: Pain neuroscience education program — 1. Types of pain (peripherical and central pain)
  2. Pain as information.
  3. Benign and harmful pain
  4. Psychological factors and pain in sport (Injuries, catastrophizing and pain)
  Arms: Intervention group
Behavioral: Self-care education program — 1. The importance of resting
  2. Nutritional habits
  3. Recovery techniques for athletes
  4. Principles of stretching, strengthening and endurance training
  Arms: Control group

SUMMARY:
This study is designed to evaluate the effects of a pain neuroscience education program in pain perception, wellness and pain catastrophizing of youth athletes. For this, an experimental study with an intervention group (IG) and a control group (CG) is designed. During 12 weeks of the 2022-2023 season, CG will receive a self-care education program, with information about health habits in the sport (rest, nutrition, body care and recovery). Meanwhile, IG will also receive a pain neuroscience education program, with information about biological, psychological and perceptual aspect of pain in the sports context. The study will be developed in the Sport High Performance Centre of Balearic Islands, from January to May. All athletes from this sports centre will be invited to participate in the study throughout an e-mail invitation from their sport regional federation. Prior to the beginning of the study, all participants will sign the inform consent. The Ethical Committee of the local university approved this study (280CER22). One week before intervention period, all athletes will be required to complete questionnaire about sociodemographic and sportive data (age, sex, and sport experience). Body mass and height will be also evaluated. Also, all the athletes will be required to complete three questionnaires about pain level, wellness and pain catastrophizing. Pain level and wellness will be evaluated prior to the start of the intervention and weekly, until finishing the intervention period. The pain catastrophizing level will be evaluated before and after the intervention period of the study. We hypothesized that those athletes who receive the pain neuroscience education program will increase wellness and decrease pain level and catastrophizing perception compared to those athletes who received a self-care educational program.

ELIGIBILITY:
Inclusion Criteria:

* to have at least 14 years old
* to have at least 2 years of experience in the sport

Exclusion Criteria:

* to have sustained an injury during the previous 6 months to start of the study
* to have sustained a surgery during the previous 12 months to start of the study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Wellness level | Change from baseline and between group differences in wellness during and after the intervention period of 12 weeks
  It is composed by seven questions about wellness, perceived effort, training volume. Wellness was assessed throughout four questions about the subjective perception of the quality of sleep, the amount of stress, the level of perceived fatigue, mood and perceived muscle damage. Each question is individually scored from 1 ("Very, very low, or very, very good") to 5 ("Very, very high, or very, very bad"), being 25 the maximal punctuation.
Pain level | Change from baseline and between group differences in pain during and after the intervention period of 12 weeks
  Pain intensity is assessed by using the Pain Visual Analog Scale (VAS, 0-10), ranging from 0 (no pain) to 10 (the worst imaginable pain). In case of pain existence, anatomical location, duration (days), sports practice affection (yes/no) were also collected
Pain catastrophizing level | Change from baseline and between group differences in pain catastrophizing after the intervention period of 12 weeks
  It is designed to evaluate the catastrophizing level of athletes throughout the Pain Catastrophism Scale (PCS). The PCS assesses catastrophic level associated to pain experience through thirteen 4-points Likert items (from 0, not at all, to 4, all the time). Apart from global Catastrophism, PCS evaluates four subscales regarding rumination, helplessness, and magnification. The maximal score is 50 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Sport High Performance Center of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Sullivan K, O'Sullivan PB, Gabbett TJ. Pain and fatigue in sport: are they so different? Br J Sports Med. 2018 May;52(9):555-556. doi: 10.1136/bjsports-2017-098159. Epub 2017 Oct 19. No abstract available. PMID 29051168
- [Background] Vicente-Mampel J, Gargallo P, Bautista IJ, Blanco-Gimenez P, de Bernardo Tejedor N, Alonso-Martin M, Martinez-Soler M, Baraja-Vegas L. Impact of Pain Neuroscience Education Program in Community Physiotherapy Context on Pain Perception and Psychosocial Variables Associated with It in Elderly Persons: A Ranzomized Controlled Trial. Int J Environ Res Public Health. 2022 Sep 20;19(19):11855. doi: 10.3390/ijerph191911855. PMID 36231171
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] Afzal Z, Mansfield CJ, Bleacher J, Briggs M. RETURN TO ADVANCED STRENGTH TRAINING AND WEIGHTLIFTING IN AN ATHLETE POST-LUMBAR DISCECTOMY UTILIZING PAIN NEUROSCIENCE EDUCATION AND PROPER PROGRESSION: RESIDENT'S CASE REPORT. Int J Sports Phys Ther. 2019 Sep;14(5):804-817. PMID 31598418
- [Background] Maguire N, Chesterton P, Ryan C. The Effect of Pain Neuroscience Education on Sports Therapy and Rehabilitation Students' Knowledge, Attitudes, and Clinical Recommendations Toward Athletes With Chronic Pain. J Sport Rehabil. 2019 Jul 1;28(5):438-443. doi: 10.1123/jsr.2017-0212. Epub 2018 Oct 15. PMID 29405811
- [Background] Hooper SL, Mackinnon LT. Monitoring overtraining in athletes. Recommendations. Sports Med. 1995 Nov;20(5):321-7. doi: 10.2165/00007256-199520050-00003. No abstract available. PMID 8571005
- [Background] Scrimshaw SV, Maher C. Responsiveness of visual analogue and McGill pain scale measures. J Manipulative Physiol Ther. 2001 Oct;24(8):501-4. doi: 10.1067/mmt.2001.118208. PMID 11677548